CLINICAL TRIAL: NCT05425953
Title: Endocrine, Metabolic, Cardiovascular and Immunological Aspects of Sex Chromosome
Brief Title: Endocrine, Metabolic, Cardiovascular and Immunological Aspects of Sex Chromosome Abnormalities in Relation to Genotype
Acronym: EMKISCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EMKI SCA
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Sex Chromosome Abnormality; Klinefelter Syndrome; Turner Syndrome; Metabolic Disease; Cardiovascular Diseases; Immunologic Disease
MeSH Terms: conditions — Sex Chromosome Aberrations; Klinefelter Syndrome; Turner Syndrome; Metabolic Diseases; Cardiovascular Diseases; Immune System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biopsies from skin, muscle, fat, urine, buccal swaps and blood will be analysed for DNA and RNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Klinefelter syndrome: Patients with 47, XXY n=60
  Interventions: Other: No intervention other than obtaining biopsies
- Turner syndrom: Patients with 45, X n=60
  Interventions: Other: No intervention other than obtaining biopsies
- 47, XXX: Patients with 47, XXX n=20
  Interventions: Other: No intervention other than obtaining biopsies
- 47, XYY: Patients with 47, XYY n=20
  Interventions: Other: No intervention other than obtaining biopsies
- Male controls: Male controls n=80
  Interventions: Other: No intervention other than obtaining biopsies
- Female controls: Female controls n=80
  Interventions: Other: No intervention other than obtaining biopsies

INTERVENTIONS:
Other: No intervention other than obtaining biopsies — Biopsies will be obtained.

SUMMARY:
Observational study of 160 patients with sex-chromosome abnormalities and 160 matched controls. Blood, fat, muscle, skin, buccal swaps, urine will be collected and analyzed for DNA, RNA and methylation patterns. The goal is to associated genotype and epigenetic changes with the phenotype of patients with sex-chromosome abnormalities.

Patients participate in questionaries, dexa-scan of bones, fibroscan of liver, ultra sound of testicles and blood will be analyzed for organ specific blood work as well as immunological and coagulation components.

DETAILED DESCRIPTION:
Background: The most prevalent SCAs are Klinefelter syndrome (KS; 47, XXY), 47,XXX, 47,XYY and Turner syndrome (TS; 45,X) with a prevalence of 85-250, 84, 98 and 50 per 100,000 liveborn boys/girls, respectively. The majority of SCAs can suffer from a range of diseases including congenital malformations, metabolic diseases, hypergonadotropic hypogonadism and infertility, autoimmune disease and psychiatric diseases. However, the genetic mechanisms causing these phenotypes are largely unexplained. The phenotypes have been suggested to arise from alterations in DNA methylation and RNA-expression. The methylome and transcriptome in peripheral blood samples from persons with KS, 47,XXX and TS have been found to be altered in comparison with controls. These genes are now starting to be found ex. SHOX, located in the pseudo autosomal region of the X and Y chromosome, escapes X-inactivation and is therefore equivalent to the number of sex chromosomes. Altered expression of SHOX in SCAs has been associated with the altered height seen in these patients.

Hypotheses:

1. The methylome and transcriptome of SCAs is altered compared to karyotypical normal female and males, and a unique methylation profile and RNA expression profile is seen for the different SCAs subgroups.
2. The methylation profile and the RNA expression profile show temporal alterations.
3. The DNA methylation profile and the RNA expression profile are tissue-specific.

3. The phenotype and the increased risk of diseases seen in patients with SCAs are associated with the altered RNA-expression and DNA methylation profile.

Materials: Blood, fat, muscle, skin, buccal swaps, urine, will be collected from 60 klinefelter, 60 Turner syndrome patient, 20: 47, XXX and 20: 47, XYY and 80 male and female matched controls.

Methods:

Analysis of DNA-methylation using Whole Genome Bisulfite Sequencing (WGBS). Genomic DNA will be bisulfite-converted and sequenced on an Illumina Novaseq System. Sequence data pre-processors of software pipeline MethylStar. Analyzed using R.

Gene expression analysis (RNA) RNA will be cleaned and sequenced with a sequence depth of 30 million reads. Processing of sequence data using FastQC (quality control), HISAT2 (mapping) and featureCounts (gene-expression). Differences in gene-expression will be analyzed in R.

The extracted biopsies will be dissociated to singular cells RNA from these singular cells will be individually sequenced. For miRNA analysis we will isolate small non-coding RNAs and analyze these by next generation sequencing. Chromatin re-modelling can be analyzed through "footprints" left by histones on DNA-strand. Mapping of footprints along the whole X-chromosome is done using a single assay with chromatin-immunoprecipitation (CHIP) in combination med deep sequencing (chIPseq).

Genotype-Phenotype association analysis with weighted correlation network analysis (WGCNA) we will uncover the patterns in which genes behave and divide them into modules where genes react dependent of each other. These modules will afterwards be associated with the clinical data, enabling identification of the "hub" genes with the strongest associations to the phenotype.

These gene-modules, and the gene expression data itself, can furthermore be included in "deep-phenotyping" using artificial intelligence Perspectives A characterization of the methylome and transcriptome from different target tissue from patients with SCAs would not just be of significance to these patients but could lead to a larger understanding of similar diseases in patients without SCAs. Using SCAs as disease models and identify changes in DNA methylation and RNA-expression related to co-morbidity such as the metabolic syndrome, congenital heart disease or psychiatric diseases could increase the understanding of these diseases in general and potentially improve treatment in other patients groups with similar diseases.

In addition, the data collection will expand our biobank and will enable future research projects about SCAs.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have the sex-chromosome abnormality

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Study population are danish participants.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Epigenetic changes relate to phenotype | 2½ years
  Epigenetic changes relate to phenotype

SECONDARY OUTCOMES:
Immunologic changes in turner syndrom | 2 years
  Patients with Turner syndrome may have altered immunological properties

CONTACTS AND LOCATIONS:
Overall Officials: Claus Gravholt, Prof, Study Director — Aarhus University Hospital
Locations (1):
- Aarhus university hospital, Aarhus, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roulot D, Degott C, Chazouilleres O, Oberti F, Cales P, Carbonell N, Benferhat S, Bresson-Hadni S, Valla D. Vascular involvement of the liver in Turner's syndrome. Hepatology. 2004 Jan;39(1):239-47. doi: 10.1002/hep.20026. PMID 14752843
- [Background] Gravholt CH, Chang S, Wallentin M, Fedder J, Moore P, Skakkebaek A. Klinefelter Syndrome: Integrating Genetics, Neuropsychology, and Endocrinology. Endocr Rev. 2018 Aug 1;39(4):389-423. doi: 10.1210/er.2017-00212. PMID 29438472
- [Background] de Vos WM, Tilg H, Van Hul M, Cani PD. Gut microbiome and health: mechanistic insights. Gut. 2022 May;71(5):1020-1032. doi: 10.1136/gutjnl-2021-326789. Epub 2022 Feb 1. PMID 35105664
- [Result] Berglund A, Viuff MH, Skakkebaek A, Chang S, Stochholm K, Gravholt CH. Changes in the cohort composition of turner syndrome and severe non-diagnosis of Klinefelter, 47,XXX and 47,XYY syndrome: a nationwide cohort study. Orphanet J Rare Dis. 2019 Jan 14;14(1):16. doi: 10.1186/s13023-018-0976-2. PMID 30642344
- [Result] Gravholt CH, Juul S, Naeraa RW, Hansen J. Prenatal and postnatal prevalence of Turner's syndrome: a registry study. BMJ. 1996 Jan 6;312(7022):16-21. doi: 10.1136/bmj.312.7022.16. PMID 8555850
- [Result] Elsheikh M, Hodgson HJ, Wass JA, Conway GS. Hormone replacement therapy may improve hepatic function in women with Turner's syndrome. Clin Endocrinol (Oxf). 2001 Aug;55(2):227-31. doi: 10.1046/j.1365-2265.2001.01321.x. PMID 11531930
- [Result] Gravholt CH, Poulsen HE, Ott P, Christiansen JS, Vilstrup H. Quantitative liver functions in Turner syndrome with and without hormone replacement therapy. Eur J Endocrinol. 2007 Jun;156(6):679-86. doi: 10.1530/EJE-07-0070. PMID 17535868
- [Result] Ahmed S, Spence JD. Sex differences in the intestinal microbiome: interactions with risk factors for atherosclerosis and cardiovascular disease. Biol Sex Differ. 2021 May 17;12(1):35. doi: 10.1186/s13293-021-00378-z. PMID 34001264
- [Result] Org E, Mehrabian M, Parks BW, Shipkova P, Liu X, Drake TA, Lusis AJ. Sex differences and hormonal effects on gut microbiota composition in mice. Gut Microbes. 2016 Jul 3;7(4):313-322. doi: 10.1080/19490976.2016.1203502. Epub 2016 Jun 29. PMID 27355107